CLINICAL TRIAL: NCT00459342
Title: Phase II Study of Dasatinib in Non Small Cell Lung Cancer
Brief Title: Dasatinib in Treating Patients With Stage IIIB, Stage IV, or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00225; NCI-2009-00225 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000538668; 2006-0593; 2006-0593 (Other: M D Anderson Cancer Center); 7798 (Other: CTEP); N01CM62202 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Non-small Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Dasatinib

ARMS (1):
- Arm I (Experimental): Patients received oral dasatinib twice daily on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — Given orally
  Other Names: BMS-354825; Sprycel

SUMMARY:
Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. This phase II trial is studying how well dasatinib works in treating patients with stage IIIB, stage IV, or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the progression-free survival at 12 weeks in patients with stage IIIB or IV or recurrent non-small cell lung cancer treated with dasatinib.

SECONDARY OBJECTIVES:

I. Determine the rate of response in patients treated with this drug. II. Examine the relationship between clinical response to this drug and epidermal growth factor receptor (EGFR) mutational status, EGFR copy number, and (phosphorylated Src) pSrc expression levels in pre-treatment tumor biopsies.

III. Determine the toxicity of this drug.

OUTLINE:

Patients received oral dasatinib twice daily on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Previously obtained paraffin-embedded tumor tissue samples are analyzed by polymerase chain reaction and fluorescent in situ hybridization (FISH) for epidermal growth factor receptor and by immunohistochemistry for pSrc expression.

ELIGIBILITY:
Inclusion Criteria:

* Platelet count >= 100,000/mm^3
* Histologically or cytologically confirmed non-small cell lung cancer meeting 1 of the following criteria:

  * Stage IV disease
  * Stage IIIB disease with pleural effusion
  * Recurrent disease after surgery or radiotherapy
* Measurable disease, defined as >= 1 lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded) >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan
* Previously treated brain metastasis allowed, provided there is no bleeding, no midline shift, no need for steroids or anti-convulsants, and no symptoms
* Must agree to obtain residual tumor tissue available from the existing diagnostic biopsy tumor tissue
* Eastern cooperative oncology group (ECOG) performance status (PS) 0-1 OR Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* White blood cell (WBC) >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and ALT =< 2.5 times ULN
* Creatinine =< 3 times ULN OR Creatinine clearance >= 60 mL/min
* No uncontrolled congestive heart failure or potentially life-threatening arrhythmia
* No angina at rest
* No neuropathy >= grade 2
* No chronic diarrhea or history of inflammatory bowel disease
* No history of pulmonary fibrosis (other than in an irradiated field)
* No other concurrent serious medical illness
* O2 saturation > 92% on room air
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions to compounds of similar chemical or biological composition to dasatinib
* No heart rate-corrected QT interval (QTc) prolongation (i.e., QTC >= 480 msec) or other significant ECG abnormalities that could lead to adverse effects if the QTc interval were prolonged
* No medical condition that impairs the ability to swallow, retain, or absorb dasatinib including, but not limited to, any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication, requirement for IV alimentation, prior surgical procedures affecting absorption, active peptic ulcer disease
* No myocardial infarction or ventricular tachyarrhythmia within the past 6 months
* left ventricular ejection fraction (LVEF) normal
* No major conduction abnormality (unless cardiac pacemaker is present)
* No ongoing or active infection
* No history of significant bleeding disorder (congenital [von Willebrand's disease] or acquired [antifactor VIII antibodies])
* No psychiatric illness or social situation that would preclude study compliance
* No prior chemotherapy or biologic therapy for recurrent or metastatic non-small cell lung cancer
* Adjuvant cytotoxic chemotherapy after surgical resection or chemotherapy with radiation for locally advanced disease (curative intent) allowed provided disease recurrence >= 3 months after completion of last chemotherapy dose
* Measurable disease must be outside the radiotherapy port OR clearly growing inside the port
* No prior radiotherapy to >= 25% of the marrow-containing skeleton
* At least 7 days since prior and no concurrent medications that are inhibitors or inducers of CYP3A4
* At least 7 days since prior and no concurrent agents with proarrhythmic potential
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies
* No concurrent antiretroviral therapy for HIV-positive patients
* No concurrent systemic antacids (H2 receptor antagonists and proton pump inhibitors)
* Locally acting antacids allowed except for 2 hours before and after dasatinib administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faye Johnson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 22, 2007 to April 20, 2009. All recruitment done at UT MD Anderson Cancer Center.
Groups:
- Dasatinib: Oral dasatinib 100 mg (two 50 mg tablets) twice daily on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dasatinib
Started | 35
Completed | 34
Not Completed | 1
Not completed — Not eligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 69 [51 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response (Complete Response (CR) or Partial Response (PR))
Description: Objective response defined as participants with Complete Response (CR) or Partial Response (PR) evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. RECIST definitions are Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started. Response measured by tumor size on computed tomography scans and by metabolic activity on positron emission tomography scans.
Time Frame: 12 weeks
Population: Of the 34 eligible study participants enrolled, four participants were not evaluable for response.
Measure: Number; unit: participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 30
participants
  Partial Remission | 1
  Stable Disease | 12
  Progressive Disease | 17

2. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death.
Time Frame: Time from start of treatment to time of progression or death, assessed at 2 months
Population: Four participants were not evaluable for response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib
Number analyzed (Participants) | 30
months | 1.36 [0.16 to 17.2]

3. Other Pre Specified Outcome: Time to Progression (TTP)
Time Frame: Time from start of treatment to time of progression or death, assessed radiographically every 6 weeks
Population: Seven patients discontinued dasatinib because of toxicity or unrelated medical problems (i.e., not progression) and are not evaluable for progression.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dasatinib
Number analyzed (Participants) | 27
days | 92 (107)

4. Other Pre Specified Outcome: Epidermal Growth Factor Receptor (EGFR) Mutational Status
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 34
participants
  EGFR mutant | 9
  EGFR wild type | 22
  EGFR not tested | 3

5. Other Pre Specified Outcome: Epidermal Growth Factor Receptor (EGFR) Copy Number
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 34
participants
  EGFR amplfied | 3
  EGFR not amplified | 17
  EGFR copy number unknown | 14

6. Other Pre Specified Outcome: Phospho-Src (pSrc) Expression
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 34
participants
  pSrc positive | 10
  pSrc negative | 11
  pSrc unknown | 13

ADVERSE EVENTS:
Time Frame: 29 weeks
Description: Treatment schedule included up to eight (8) possible 21-day (3-week) study cycles with follow up about 4-5 weeks after the last dose of Dasatinib.
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 25/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=35)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (17)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hypoxia (Blood and lymphatic system disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Thromboembolic event (Blood and lymphatic system disorders) | 2 (2)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Headache (General disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=35)
Abdominal pain (General disorders) | 2 (2)
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 3 (3)
Allergic rhinitis (Immune system disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 6 (9)
Anorexia (Metabolism and nutrition disorders) | 16 (17)
Anxiety (Psychiatric disorders) | 6 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate aminotransferase increased (Endocrine disorders) | 3 (3)
Back pain (General disorders) | 6 (6)
Bladder infection (Renal and urinary disorders) | 1 (1)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (25)
Depression (Psychiatric disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 15 (17)
Dizziness (Nervous system disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dysgeusia (Musculoskeletal and connective tissue disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 (32)
Edema face (Skin and subcutaneous tissue disorders) | 4 (5)
Edema limbs (Skin and subcutaneous tissue disorders) | 3 (3)
Epistaxis (General disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 28 (39)
Fever (Infections and infestations) | 3 (5)
Flatulence (Gastrointestinal disorders) | 2 (2)
Flushing (Skin and subcutaneous tissue disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 3 (3)
Headache (General disorders) | 9 (9)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 5 (5)
Hypoalbuminemia (Endocrine disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypothyroidism (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Blood and lymphatic system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 7 (8)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 11 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 21 (22)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
Nipple deformity (Reproductive system and breast disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1)
Pelvic pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 18 (26)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (9)
Respiratory, thoracic and mediastinal disorders - (Other) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tracheal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Voice alteration (Nervous system disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (7)
Weight loss (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less